CLINICAL TRIAL: NCT02625688
Title: The Risk of Hyperbilirubinemia in Term Newborns After Placental Transfusion: A Randomized-blinded Controlled Trial
Brief Title: The Risk of Hyperbilirubinemia in Term Newborns After Placental Transfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Joanna Seliga-Siwecka, Assistant, Princess Anna Mazowiecka Hospital, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1/2013
Record Dates: First submitted 2015-11-26; First posted 2015-12-09 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Jaundice Neonatal
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early cord clamping (Placebo Comparator): Cord clamping will be applied after 30 seconds post delivery.
  Interventions: Other: Early cord clamping
- Delayed cord clamping (Active Comparator): Cord clamping will be applied after 3 minutes post delivery.
  Interventions: Other: Delayed cord clamping
- Cord milking (Active Comparator): The baby will be placed below the level of the placenta, between the mother's thighs (during a vaginal delivery) or at the side of the mother swaddled in sterile towels (during a caesarian delivery).
  Interventions: Other: Cord milking

INTERVENTIONS:
Other: Delayed cord clamping — We have decided to delay cord clamping in the intervention group to 3 minutes and place the baby 10 cm above the placental, as it seems most efficient based on the available literature. At all births (spontaneous vaginal deliveries and caesarian sections) a member of the recruitment team will be present. He will inform the midwife or obstetrician about the allocated intervention and measure the time from the delivery of the shoulders to the cord clamping.
  Arms: Delayed cord clamping
Other: Cord milking — If cord milking will be the allocated intervention, the recruiter will supervise the midwife, or obstetrician preforming the procedure, and count out loud the number of times the cord has been milked. During vaginal deliveries midwifes will be asked to maintain the infant at least 10 cm above the uterus until the cord is clamped. In case of caesarian sections the baby will be placed on the mother's laps and swaddled in sterile towels to prevent heat loss.
  Arms: Cord milking
Other: Early cord clamping — We have decided to clamp the cord in the early intervention group at 30 seconds and place the baby 10 cm above the placental, as it seems most efficient based on the available literature. At all births (spontaneous vaginal deliveries and caesarian sections) a member of the recruitment team will be present. He will inform the midwife or obstetrician about the allocated intervention and measure the time from the delivery of the shoulders to the cord clamping.
  Arms: Early cord clamping

SUMMARY:
Delayed cord clamping (DCC) has been a subject of extensive research for the last couple of years. Based on published data, numerous neonatal benefits have been suggested such as increased hemoglobin and ferritin levels both at birth and longer term. Available systematic reviews of DCC versus early cord clamping (ECC) reveal that it may also contribute to other neonatal outcomes including polycythemia and hyperbilirubinemia.

A review published nearly 10 years ago regarding late umbilical cord clamping revealed only 4 studies which as a second objective assessed whether the time of cord clamping was associated with an increased risk of polycythemia and hyperbilirubinemia during the first week of life. Two studies reported that neonates with DCC had bilirubin levels >15 mg/dl. No information is provided on what hour of life the bilirubin levels were measured exactly.

In this randomized control study the investigators would like to determine if delayed cord clamping or cord milking during labor increases the risk of hyperbilirubinaemia (requiring phototherapy) in term infants.

DETAILED DESCRIPTION:
The investigators feel that published results regarding 'jaundice" and "jaundice needing phototherapy' (associated with DCC) may be misleading.

First, no information is offered about how "clinical jaundice "was assessed on examination. The absence of jaundice is not an indication of the absence of hyperbilirubinemia. Estimation of the degree of hyperbilirubinemia based solely on clinical examination can lead to errors. The absence or the severity of jaundice is not predictive of subsequent severe hyperbilirubinemia. A recent study revealed that the nurses' predischarge assessment of jaundice extent was only moderately correlated with bilirubin concentration and was similar in black and nonblack infants.

A review published nearly 10 years ago regarding late umbilical cord clamping revealed only 4 studies which as a secondary objective which assessed whether the time of cord clamping was associated with an increased risk of polycythemia and hyperbilirubinemia during the first week of life. Two studies reported that neonates with DCC had bilirubin levels >15 mg/dl. No information is provided on what hour of life the bilirubin levels were measured exactly.

Secondly, guidelines to treat jaundice have changed over time and none of the studies mention what threshold was used for administering phototherapy. No information is given if, staff responsible for phototherapy administration was blinded to the type of cord clamping intervention. Potential confounders such as isoimmune hemolytic disease, symptoms of sepsis (significant lethargy, temperature instability), asphyxia, G6PD, acidosis, albumin <3 g/L were not included in the analysis. Also another important factor such feeding policy at the time of bilirubin measurement wasn't mentioned in neither of the studies.

The presence of all mentioned above confounders in available studies has lead the investigators to conduct a blinded randomized trial.

Postnatal hyperbilirubinemia is universal and manifests as newborn jaundice in over 60-80% of all newborns. If left untreated hyperbilirubinemia may progress to excessive levels that can be associated with evident bilirubin neurotoxicity. Jaundice is the most common clinical diagnosis in neonatal medicine. Elevated bilirubin concentrations may occur due to increased bilirubin production (breakdown of heme moiety of hemoglobin) and/or delayed bilirubin elimination (hepatic and intestinal) as well as by a unique neonatal phenomenon of enterohepatic reabsorption of bilirubin.

Studies have shown that late cord clamping benefits expand beyond the neonatal period. A meta -analyses estimated a significant 47% reduction in the risk of anemia and 33% reduction in risk of having deficient iron stores at ages 2 to 3 months in the delayed cord clamping group. These pooled results are based on two small studies, and despite a significant number of patients lost to follow up (40%), these results agree with a large randomized trial.

It is important to understand whether evidence based benefits of DCC (such as increase of hemoglobin, improved iron status, and decreased risk of infant anemia) may also contribute to less favorable neonatal outcomes. This trial will aim to assess if delayed cord clamping truly increases the risk of hyperbilirubinaemia requiring phototherapy or even exchange transfusion.

Dose selection:

The total feto-placental blood volume is about 120 ml/kg of fetal weight. At birth, the distribution of blood between fetus and placenta is roughly at a ratio of 2:1. Increasing placental transfusion to at least three minutes leads to a larger infant blood volume (ratio 5:1).The rate of placental transfusion is markedly influenced by the position of the delivered infant. From at least 10 cm above to at least 10 cm below the level of the placenta, infants receive the maximum possible amount after at least three minutes of birth .

The randomized and quasi-randomized controlled trials that studied delayed cord clamping in vaginally born, healthy, term infants differed in clamping time and infant position before clamping and there is still no consensus about the time required for a sufficient amount of blood to be transfused from the placenta to the baby. The above mentioned trials showed that placental-neonate blood flow significantly increases after DCC by showing higher packed cell volume or hemoglobin concentration in the first 24 hours after birth compared with immediate clamping.

To test the hypothesis, investigators have decided to delay cord clamping in the intervention group to 3 minutes and place the baby 10 cm above the placental, as it seems most efficient based on the available literature. At all births (spontaneous vaginal deliveries and caesarian sections) a member of the recruitment team will be present. He will inform the midwife or obstetrician about the allocated intervention and measure the time from the delivery of the shoulders to the cord clamping. If cord milking will be the allocated intervention, the recruiter will supervise the midwife, or obstetrician preforming the procedure, and count out loud the number of times the cord has been milked. During vaginal deliveries midwifes will be asked to maintain the infant at least 10 cm above the uterus until the cord is clamped. In case of caesarian sections the baby will be placed on the mother's laps and swaddled in sterile towels to prevent heat loss. In the early cord clamping group, the recruiter will inform the midwife or obstetrician when 30 seconds have passed. In the delayed clamping group, the recruiter will inform the midwife or obstetrician after 3 minutes.

If cord milking will be applied the baby will be placed below the level of the placenta, between the mother's thighs (during a vaginal delivery) or at the side of the mother swaddled in sterile towels (during a caesarian delivery). Based on available literature, before starting the trial investigators piloted this procedure[13]. They checked that about two thirds of the umbilical cord will be present for milking both during a vaginal and caesarian delivery. If the cord was milked once we were able to transfer approximately 10 ml of blood to the neonate. Following this, and under the assumption that the cord vein will be rapidly refilling itself, investigators assume that milking the cord four times will give us 40 ml of blood [13]. A member of the delivery team (vaginal delivery) or operating team (caesarian delivery) will hold the cord at the level of the introitus or cesarean wound, and milk the cord four times towards the neonate counting out loud. The cord will be clamped after the forth milking.

Choice of comparator In spite of available studies which advocate for delayed cord clamping, it is still infrequently used in labor wards throughout the world[28]. According to the new guidelines early cord clamping-ECC is defined as cord clamping at less than 60 seconds after the delivery. The available meta-analyses comparing early versus late cord clamping include studies which significantly vary in defining ECC. The majority of trials define ECC as clamping within the first 10 seconds, other describe ECC as immediate clamping. Only one trial extended ECC to be as long as 60 seconds.

The new 2010 ILCOR (International Liaison Committee on Resuscitation) guidelines advocate for DDC, stating that cord clamping should be delayed for at least 1 min from the complete delivery of the baby. Investigators have chosen this definition, as the ILCOR committee provides an international consensus and evidence based guidelines on emergency care, which are widely accepted among neonatologist throughout the world.

ECC is part of active management of labour. Active management usually involves the clinician intervening in the process through three interrelated processes: the administration of a prophylactic uterotonic drug; cord clamping and cutting at ≤60 seconds after delivery; and controlled traction of the umbilical cord. These interventions are aimed at reduction in the risk of postpartum haemorrhage. However, ECC eliminates the possibility of additional blood flowing from the placenta to the newborn, and deprives the baby from numerous profits such as receiving extra amounts of iron. This potential additional amount of iron prevents iron deficiency during the first year of life in infants born with delayed cord clamping.

Research Hypothesis Neither delayed cord clamping nor cord milking during labor does not increase significantly the risk of hyperbilirubinaemia in comparison to early cord clamping.

Description of trial design The trail is designed as a randomized controlled, observer blinded trial with 3 parallel groups and a primary endpoint of hyperbilirubinemia requiring phototherapy. Randomization will be performed as block randomization with a 1:1:1 allocation. The experiment is designed to demonstrate non-inferiority of delayed cord clamping and cord milking group in comparison to early cord clamping group regarding the incidence of bilirubinemia treated with phototherapy in neonates.

Description of study settings The study will be carried out in the Princess Anne's Hospital in Warsaw, Poland. This is a level III teaching hospital with approximately 3500 (1000 < 37 weeks of gestation) deliveries per year and 63 neonatal beds. It is also a referral center for gestational and pre-gestational diabetes as well as pregnancy induced hypertension. Having access to high risk mothers will augment the population of small for gestation infants (SGA), and infants of diabetic mothers (IDM) in the study. SGA and IDM have an increased risk for hyperbilirubinemia, thus the presence of the above patients will improve the generalizability of the study population. The local protocol on cord clamping has not yet been adjusted to the new ILCOR guidelines, but labour ward staff are willing to implement new procedures. This should improve trail recruitment and adherence.

ELIGIBILITY:
Inclusion Criteria

All maternal-fetal dyads must comply with all of the following at randomization:

* Term delivery between 37 -42 weeks of gestation (estimated by ultrasound).
* Signed parental consent.
* Singleton delivery.
* Nonsmoking mothers.
* Mothers willing to return for follow up visits.
* Declaration of breastfeeding for at least six months.

Exclusion Criteria The following maternal - fetal dyads will be excluded

1. Preterm delivery < 37 weeks of gestation (estimated by ultrasound).
2. Isoimmune hemolytic disease.
3. Sepsis.
4. Maternal Gilbert syndrome.
5. Birth asphyxia.
6. Serious maternal hemorrhage during delivery.
7. Major congenital abnormalities.
8. Need for early cord clamping (tight nuchal cord, need for resuscitation).
9. Participation in another trial.

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The number of patients with hyperbilirubinemia requiring phototherapy or exchange transfusion. | 14 days of life
  Infants requiring phototherapy or exchange transfusion will be evaluated according to the AAP guidelines. The above evidence based guidelines describe the management of neonatal hyperbilirubinaemia in newborns above 35 weeks of gestation. Serum bilirubin levels will be interpreted according to the baby's age in hours. Physicians assessing the infant and prescribing phototherapy will be blinded to treatment.

SECONDARY OUTCOMES:
The number of patients with polycythemia defined as a hematocrit > 65%. | 48-72 hours of life.
  Hematocrit levels peak at about 2 hours of age, and gradually stabilize during the following 12-24 hours. To avoid bias and minimalize the amount of needle pricks we have chosen to combine serum bilirubin and hematological measurements to the minimal amount of samples .
The number of patients with symptomatic polycythemia (hematocrit > 75%), and non - symptomatic polycythemia (hematocrit >80%). | 48-72 hours of life
  Symptomatic polycythemia (hematocrit > 75%), non - symptomatic polycythemia (hematocrit >80%) requiring exchange transfusion during the 48-72 hours of life
The number of patients with symptomatic polycythemia defined as lethargy, plethora, jitteriness, tachycardia, tachypnea | 48-72 hours of life
The number of patients with congenital anemia | at birth
  cord Hb <12.5 g/dL

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Seliga-Siwecka, MD Phd, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw, Poland

REFERENCES:
- [Background] Bhutani VK, Gourley GR, Adler S, Kreamer B, Dalin C, Johnson LH. Noninvasive measurement of total serum bilirubin in a multiracial predischarge newborn population to assess the risk of severe hyperbilirubinemia. Pediatrics. 2000 Aug;106(2):E17. doi: 10.1542/peds.106.2.e17. PMID 10920173
- [Background] Rubaltelli FF, Gourley GR, Loskamp N, Modi N, Roth-Kleiner M, Sender A, Vert P. Transcutaneous bilirubin measurement: a multicenter evaluation of a new device. Pediatrics. 2001 Jun;107(6):1264-71. doi: 10.1542/peds.107.6.1264. PMID 11389241
- [Background] Bhutani VK, Johnson L, Sivieri EM. Predictive ability of a predischarge hour-specific serum bilirubin for subsequent significant hyperbilirubinemia in healthy term and near-term newborns. Pediatrics. 1999 Jan;103(1):6-14. doi: 10.1542/peds.103.1.6. PMID 9917432
- [Background] Keren R, Tremont K, Luan X, Cnaan A. Visual assessment of jaundice in term and late preterm infants. Arch Dis Child Fetal Neonatal Ed. 2009 Sep;94(5):F317-22. doi: 10.1136/adc.2008.150714. Epub 2009 Mar 22. PMID 19307221
- [Background] McDonald SJ, Middleton P. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD004074. doi: 10.1002/14651858.CD004074.pub2. PMID 18425897
- [Background] Gupta R, Ramji S. Effect of delayed cord clamping on iron stores in infants born to anemic mothers: a randomized controlled trial. Indian Pediatr. 2002 Feb;39(2):130-5. PMID 11867842
- [Background] Ceriani, R.J., Ferreira C. P. , M. A., Effect of Timing of Cord Clamping on Postnatal Hematocrit Values and Clinical Outcome in Term Infants. A Randomized, Controlled Trial. Pediatr Res, 2005. 57(6): p. 922-922.
- [Background] Bhutani, V.K., Screening for severe neonatal hyperbilirubinemia. Pediatric Health, 2009. 3(4): p. 369-379.